CLINICAL TRIAL: NCT05671575
Title: A Study of The Knowledge and Attitude Towards Epilepsy Among Close Relatives of People With Epilepsy and Their Impact on The Patient's Quality of Life
Brief Title: Study The Knowledge and Attitude Towards Epilepsy Among Relatives of People With Epilepsy and Their Impact on The Patient's Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mohamed Adel Abdellah (Other)
Responsible Party: Sponsor-Investigator, Mohamed Adel Abdellah, neuropsychiatry resident, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-22-11-05
Record Dates: First submitted 2022-11-27; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; Knowledge and Attitude; Quality of life
MeSH Terms: conditions — Epilepsy; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire about Epilepsy — After obtaining informed consent, a structured questionnaire will be administered to the accompanying relative. The questionnaire consists of 5 sections: participants socio-demographic characteristics, patient demographic and clinical characteristics, participants knowledge about epilepsy including sources of knowledge and management of an acute seizure, general attitudes, and behaviors towards the People with epilepsy, Stigma scale of epilepsy.[14], and Quality of life in epilepsy-10 inventory (QOLIE-10) as the main data collection tool as regard quality of life of patients with epilepsy.

SUMMARY:
Epilepsy is a common neurological condition that affects personal and familial behavior and social support . About 50 million people worldwide suffer from epilepsy and the prevalence of active epilepsy in developing countries is 5 to 10 per 100 persons . Individuals with epilepsy may suffer from psychological issues such as depression, anxiety, and psychosis . Accordingly, living with a person with epilepsy will provide some challenges, particularly at home. Studies have reported that relatives of people with epilepsy have an increased risk of anxiety. Epilepsy can inflict an enormous burden on both the people with epilepsy (PWE) and their family caregivers, decreasing their quality of life and daily efficiency.

ELIGIBILITY:
Inclusion Criteria:

* The participants Will be the close relatives of people with epilepsy who had a close relationship with the patient and living in the same house. The respondents will include the mothers, fathers, brothers, sisters, or the husband/wife, sons of patients.

The patients will be patients diagnosed of epilepsy for at least 6 months, who were using antiepileptic drugs.

Exclusion Criteria:

* The Relatives not living in the same house or not in direct contact with the patients or younger than 16 years old will be excluded from the study.

The persons who had major medical or mental health problems other than epilepsy that would affect QOL will be excluded.

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: participants Will be the close relatives of people with epilepsy who had a close relationship with the patient and living in the same house. The respondents will include the mothers, fathers, brothers, sisters, or the husband/wife, sons of patients.
  The patients will be patients diagnosed of epilepsy for at least 6 months, who were using antiepileptic drugs.
  The patients will be patients diagnosed of epilepsy for at least 6 months, who were using antiepileptic drugs.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge and attitudes toward epilepsy among close Relatives of people with Epilepsy. | 1 year
  This study will be conducted to assess the degree of knowledge and attitudes toward epilepsy among close Relatives of people with Epilepsy. A structured questionnaire will be administered to the accompanying relative. The questionnaire will assess this knowledge and the sources that close relatives obtain this knowledge from, including general attitude towards the People with epilepsy, and contains section that assess sigma about epilepsy using Stigma scale of epilepsy.
Quality of life of people with epilepsy. | 1 year
  We will use the Quality of life in epilepsy-10 inventory (QOLIE-10) as the main collection tool as regard quality of life of people with epilepsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekeh BC, Ekrikpo UE. The Knowledge, Attitude, and Perception towards Epilepsy amongst Medical Students in Uyo, Southern Nigeria. Adv Med. 2015;2015:876135. doi: 10.1155/2015/876135. Epub 2015 Mar 31. PMID 26556558
- [Background] Ohaeri JU, Awadalla AW, Farah AA. Quality of life in people with epilepsy and their family caregivers. An Arab experience using the short version of the World Health Organization quality of life instrument. Saudi Med J. 2009 Oct;30(10):1328-35. PMID 19838443
- [Background] Mollaoglu M, Mollaoglu M, Durna Z. Validity and Reliability of the Quality of Life in Epilepsy Inventory (QOLIE-10) For Turkey. Noro Psikiyatr Ars. 2017 Sep;54(3):239-243. doi: 10.5152/npa.2016.13809. Epub 2017 Jan 12. PMID 29033636
- [Background] Bener A, al-Marzooqi FH, Sztriha L. Public awareness and attitudes towards epilepsy in the United Arab Emirates. Seizure. 1998 Jun;7(3):219-22. doi: 10.1016/s1059-1311(98)80039-3. PMID 9700835
- [Background] Wheless JW. Intractable epilepsy: A survey of patients and caregivers. Epilepsy Behav. 2006 Jun;8(4):756-64. doi: 10.1016/j.yebeh.2006.03.010. Epub 2006 May 3. PMID 16675306